CLINICAL TRIAL: NCT03761342
Title: Multiphase Evaluation of Healthier Choice Symbol (HCS) Logo: Aim 4. A Randomized Controlled Trial Evaluating the Relative Effectiveness of Two Front-of-pack Nutrition Labels
Brief Title: Evaluating the Relative Effectiveness of Two Front-of-pack Nutrition Labels
Acronym: NUSMart NM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke-NUS Graduate Medical School (Other)
Collaborators: National Medical Research Council (NMRC), Singapore (Other Government)
Responsible Party: Principal Investigator, Eric A. Finkelstein, Professor, Duke-NUS Graduate Medical School
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: NUSMart NM
Record Dates: First submitted 2018-11-28; First posted 2018-12-03 (Actual); Last update posted 2019-01-03 (Actual); Status verified 2019-01

CONDITIONS: Diet Habit; Diet Modification; Food Selection; Food Preferences; Nutrition Poor
Keywords: Front-of-pack label; Nutrition label; Diet Quality; Online grocery store; Diet
MeSH Terms: conditions — Feeding Behavior; Food Preferences; Malnutrition

STUDY DESIGN:
Who Masked: Participant
Masking Description: While participants will be made aware that there are different versions of NUSMart, the exact details of the arms will not be revealed to ensure validity of results. It will be deleterious to the study to reveal the differences between study arms as that would likely confound participant responses. Since there are 3 shopping conditions (unknown to participants), each participant will be randomly assigned at baseline to 1 of 6 groups that vary the sequence of shopping conditions and which shops will result in an actual food delivery.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): A control arm that mirrors a traditional web-grocery store with no but with no FOP labels.
- Multiple Traffic Light Labels (Experimental): Similar to Arm 1, with Multiple Traffic Light labels displayed on all products FOP. A 60-second introductory video briefly explaining the MTL scheme will be shown before each shop in this Arm.
  Interventions: Behavioral: Multiple Traffic Light Label
- Nutri-Score (Experimental): Similar to Arm 2, with Nutri-Score labels instead of MTL labels displayed on all products FOP. A 60-second introductory video briefly explaining the NS scheme will be shown to shoppers in this condition.
  Interventions: Behavioral: Nutri-Score Label

INTERVENTIONS:
Behavioral: Multiple Traffic Light Label — The United Kingdom's Multiple Traffic Light label has repeatedly demonstrated effectiveness and has been widely implemented in Europe. The label shows how much calories, fats, saturated fats, sugar and salt are present in a product, with associated traffic light signals for high (red), medium (amber) and low (green) percentages for each attribute.
  Arms: Multiple Traffic Light Labels
Behavioral: Nutri-Score Label — In late 2017, France began voluntary implementation of one FOP label, termed Nutri-Score, adapted from its predecessor, the 5-colour Nutrition Label. Consumer acceptability and understanding of the NS label has been demonstrated in several studies. It provides a letter score as a composite grade of a product's nutrition quality from A (best) to E (worst).
  Arms: Nutri-Score

SUMMARY:
In efforts to promote a healthy diet, the Singapore Health Promotion Board (HPB) has attempted to use Front-of-Pack (FOP) labelling to supplement traditional nutrition labelling. The Healthier Choice Symbol (HCS) identifies food items within a specific category of foods as healthier choices. The original logos were enhanced to include additional information focusing on particular macronutrients, taking one of two themes; it either indicates that a product contains more of a healthier ingredient, or less of a less healthy ingredient.

However, there is a lack of scientific evidence on the role of the existing symbols in assisting consumers make healthier food purchasing decisions. Thus far, studies have established that the United Kingdom's Multiple Traffic Lights (MTL) label, and the new French Nutri-Score (NS) label, are amongst the top performers. However, there is little consensus on which is the most effective FOP label to promote diet quality. Thus, the investigators propose to conduct the following:

Use a three arm randomized controlled trial (RCT) and an experimental fully functional web-based grocery store to test two competing approaches of front-of-pack (FOP) labelling on measures of diet quality: 1) United Kingdom's Multiple Traffic Lights label (MTL) or 2) France's Nutri-Score (NS) labelling scheme.

The investigators hypothesize that diet quality as measured by the Alternative Healthy Eating Index (AHEI-2010) (primary outcome) will be highest in the NS arm, followed by MTL, and lowest in the no logo control arm.

DETAILED DESCRIPTION:
Research Aims & hypotheses:

To use a three arm randomized controlled trial (RCT), and an experimental online grocery store developed by the team, to test two competing approaches of front-of-pack (FOP) nutrition labelling on measures of diet quality: 1) Multiple Traffic Lights (MTL) and 2) Nutri-Score (NS).

All participants will experience three different shopping conditions:

1. Arm 1: A control arm that mirrors a traditional web-grocery store with no HCS or other FOP labels.
2. Arm 2: Similar to Arm 1, with additional MTL labels displayed on all products FOP. A 60-second introductory video briefly explaining the MTL scheme will be shown before participants shop as they are assumed not to have pre-existing knowledge of the label.
3. Arm 3: Similar to Arm 2, with Nutri-Score labels instead of MTL labels displayed on all products FOP. As with the MTL, a 60-second introductory video briefly explaining the NS scheme will be shown before participants shop.

The investigators hypothesize the following:

Primary Aim: Diet quality as measured by Alternative Healthy Eating Index Scores (AHEI-2010) will be highest (best) in Arm 3, followed by Arms 2 and 1 (worst).

The investigators further hypothesize a similar ordering (Arm 3 best and Arm 1 worst) for the following secondary outcomes:

Total and per serving values of the following:

1. Energy (kCal)
2. Sugar (g)
3. Total fat (g)
4. Saturated fat (g)
5. Sodium (g)
6. Fiber (g)
7. Protein (g) And
8. Average Nutri-Score across all products purchased where A=5 and E=1, and
9. Cost per calorie and per shopping trip.

The investigators will test these hypotheses in total, and separately for foods and beverages given Singapore's focus on reducing intake of sugar-sweetened beverages. The investigators will also test whether the impact of FOP labelling is moderated by mood and level of hunger at the time of purchase, and by education or income level.

ELIGIBILITY:
Inclusion Criteria:

* Singapore resident
* Aged 21 years or older.
* Existing registered RedMart customer.

Exclusion Criteria:

* Non-Singapore Resident.
* Less than 21 years old.
* Not an existing registered RedMart customer.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2018-07-31 (Actual); Primary Completion 2018-12-03 (Actual); Study Completion 2018-12-03 (Actual)

PRIMARY OUTCOMES:
Diet Quality per shopping trip | Once a week for three weeks
  Diet quality per shopping trip, as measured by an index of diet quality, the Alternative Healthy Eating Index (AHEI-2010). The Alternate Healthy Eating Index-2010 (AHEI-2010) is an updated measure of diet quality from the original Alternate Healthy Eating Index. It was constructed based on foods and nutrients predictive of chronic disease risk that incorporates current scientific evidence on diet and health. All AHEI-2010 components are scored from 0 (worst) to 10 (best), for a total of 11 components. The total AHEI-2010 score ranges from 0 (nonadherence) to 110 (perfect adherence). Higher scores on the AHEI-2010 are strongly associated with lower risk of major chronic disease as well as risk of CVD, diabetes, heart failure, colorectal and estrogen-receptor-negative breast cancer, and total and cardiovascular mortality.

SECONDARY OUTCOMES:
Total Energy in kilocalories | Once a week for three weeks
  Total Energy (kCal)
Total Sugar in grams | Once a week for three weeks
  Total Sugar (g)
Total fat in grams | Once a week for three weeks
  Total Fat (g)
Saturated fat in grams | Once a week for three weeks
  Saturated Fat (g)
Sodium in milligrams | Once a week for three weeks
  Sodium (mg)
Fiber in grams | Once a week for three weeks
  Fiber (g)
Protein in grams | Once a week for three weeks
  Protein (g)
Energy per serving in kilocalories per serving | Once a week for three weeks
  Energy per serving (kCal per serving)
Sugar per serving in grams per serving | Once a week for three weeks
  Sugar per serving (g per serving)
Total fat per serving in grams per serving | Once a week for three weeks
  Total fat per serving (g per serving)
Saturated fat per serving in grams per serving | Once a week for three weeks
  Saturated fat per serving (g per serving)
Sodium per serving in milligrams per serving | Once a week for three weeks
  Sodium per serving (mg per serving)
Fiber per serving in grams per serving | Once a week for three weeks
  Fiber per serving (g per serving)
Protein per serving in grams per serving | Once a week for three weeks
  Protein per serving (g per serving)
Average Nutri-Score across all products purchased | Once a week for three weeks
  The Nutri-Score label was developed by the Equipe de Recherche en Epidémiologie Nutritionnelle (EREN) research team based on the British Food Standards Agency nutrient profiling system, and presents the overall nutritional quality for each food and beverage on a five-point color-coded scale from A is green (best) to E in red (worst). Average Nutri-Score across all products purchased is recoded to a score of A=5, B=4, C=3, D=2 and E=1. Maximum possible score is 5 (all A) and the lowest possible score is 1 (all E). A higher score represents higher nutritional quality.
Cost per calorie in dollars per kilocalorie | Once a week for three weeks
  Cost per calorie is calculated as total spend divided by total kilocalories ($ per kCal)
Total spend in dollars | Once a week for three weeks
  Total spend ($)

CONTACTS AND LOCATIONS:
Locations (1):
- Duke-NUS Medical School, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No